CLINICAL TRIAL: NCT04413903
Title: The Effect of Different Mechanical Ventilator Modes on Optic Nerve Diameter and Cognitive Functions in Laporoscopic Cholecystectomy Operations
Brief Title: the Effect of Different Mechanical Ventilation Modes on Optic Nerve Diameter and Conscious Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Umran Karaca, Principle İnvestigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-17/23
Record Dates: First submitted 2020-03-10; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Mechanical Ventilation
Keywords: Optic Nerve Sheath Diameter,; Minimental test

STUDY DESIGN:
Intervention Model Description: ASA I-II 60 patients aged 18-65 years undergoing laparoscopic cholecystectomy surgery according to mechanical ventilator mode; Group P (n: 30) Pressure controlled ventilation was randomly divided into Group V (n: 30) volume controlled 50% air, PEEP 5 to 8ml / kg tidal volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pressure controlled ventilation, Volum controlled ventilation (Active Comparator): Undergoing laparoscopic cholecystectomy surgery according to mechanical ventilator mode; Group P (n: 30) Pressure controlled ventilation was randomly divided into Group V (n: 30) volume controlled ventilation settings were adjusted to be 50% O2- 50% air, 8ml / kg TV (tidal volume) and PEEP 5.
  Interventions: Procedure: The Effect of Different Mechanical Ventilator Modes on Optic Nerve Diameter and Cognitive Functions in Laporoscopic Cholecystectomy Operations
- Optic Nerve Sheath Diameter (Active Comparator): In optic nerve diameter measurements; A layer of water-soluble sterile gel was applied to the closed upper eyelid. The linear 10-5 MHz ultrasound probe was carefully placed on the upper eyelid over the gel. The entrance of the optic nerve to the orbital globe in 2D mode was displayed on the monitor without applying too much pressure. After finding the optimal contrast between the retrobulbar echogenic fat tissue and vertical hypoechoic band 23, the diameter of the optic nerve sheath was measured 3 mm behind the optic disc using an electronic caliper.
  Interventions: Procedure: The Effect of Different Mechanical Ventilator Modes on Optic Nerve Diameter and Cognitive Functions in Laporoscopic Cholecystectomy Operations

INTERVENTIONS:
Procedure: The Effect of Different Mechanical Ventilator Modes on Optic Nerve Diameter and Cognitive Functions in Laporoscopic Cholecystectomy Operations — The Effect of Different Mechanical Ventilator Modes on Optic Nerve Diameter and Cognitive Functions in Laporoscopic Cholecystectomy Operations

SUMMARY:
During surgery, researchers use different methods in respiratory equipment. In the study researchers examine the effects of these methods on intraocular pressure changes by looking at the intraocular nerve diameter. Then look at the effects of these effects on patients conscious functions by asking some questions.

DETAILED DESCRIPTION:
According to the mechanical ventilator application to be applied to the patients; Group P (n: 30) pressure controlled ventilation (PCV), Group V (n: 30) volume controlled ventilation (VCV) are randomly assigned to two groups. General anesthesia will be applied to all patients. Mechanical ventilation settings will be able to 8ml / kg TV (tidal volume). Demographic data (age, gender, weight, height) of patients, duration of surgery and peroperative complications will be recorded choosen time intervals.T0: awake, T1: 5th min after induction, T2: Gas insufflation start in supine position, T3: Maximum gas pressure is reached in reverse trendelenburg position, T4:Before extubation. SAB, DAB, OAB, KAH, SpO2, Ppeek, PEEP, EtCO2, optic nerve diameter will be recorded at same times. Cognitive function test will be performed at postoperative 24th hour for comparing the first awaken routin MMDT (Mini Mental Status Detection) scale. The same test will be repeated for patients who are called for routine general surgery outpatient control 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II
* 18-65 years old

Exclusion Criteria:

* Unable to cooperate
* Presence of eye disease (detachment, retinapathy, glaucoma)
* Presence of a previous eye operation
* Those with symptoms of KIBAS (intracranial pressure increase syndrome) (Intracranial lesion, previous cerebrovascular diseases)
* BMI (body mass index> 40 kg / m2
* Obstructive and restrictive lung disease
* Pulmonary Hypertension
* Congestive Heart Failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Optic nerve sheath diameter (milimeter) | 2 hours operation time
  Optic nerve sheath diameter; It was measured from the optic nerve sheath 3 mm behind the optic disc from the closed upper eyelid. T0: Awake, T1: 5th minute after induction, T2: Gas insufflation start in supine position, T3: Maximum gas pressure is reached in reverse trendelenburg position, T4: Before extubation in supine position. A typical optic nerve sheath is generally less than 5 mm in diameter and diameters greater than 5.5 mm predict an ICP of >20 cmH2O .
Cognitive Function | 3 months after surgery
  Cognitive function test with Mini Mental Conditioning Scale was performed to the patients before the anesthesia induction and 3 months after the surgery . Mini Mental Scale points are between 0 and 30.

SECONDARY OUTCOMES:
Peroperative Complications | 2 hours operation time
  Complications during the surgery (hypercapnia, hypotension,hypertension,rythm disorder) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Onur, MD, Study Chair — BYIEAH; Korgun Okmen, MD, Study Chair — BYIEAH; Serkan Terkancıoglu, MD, Study Chair — BYIEAH; Gorkem Cevik, MD, Study Chair — BYIEAH
Locations (1):
- University of Health Sciences Bursa Yüksek İhtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karaca U, Onur T, Okmen K, Terkanlioglu S, Cevik G, Ata F. Effect of Various Modes of Mechanical Ventilation in Laparoscopic Cholecystectomies on Optic Nerve Sheath Diameter and Cognitive Functions. J Laparoendosc Adv Surg Tech A. 2021 Jul;31(7):808-813. doi: 10.1089/lap.2020.0866. Epub 2020 Dec 11. PMID 33306936